CLINICAL TRIAL: NCT04675723
Title: The Role of Mucosal Microbiome in Recurrence of Clostridioides Difficile Infection
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Purna C. Kashyap, MBBS, Principal Investigator, Mayo Clinic
Other Study IDs: 19-005227
Record Dates: First submitted 2020-12-09; First posted 2020-12-19 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Clostridioides Difficile Infection
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is being done to identify types of bacteria associated with the lining of the large intestine in people who have recently been treated for C. difficile infection to determine if there are features associated with recurrent disease.

DETAILED DESCRIPTION:
Patients who have recently been diagnosed with C. difficile infection and completed treatment will be enrolled to undergo evaluation of the colonic mucosa via sigmoid biopsies. Participants will also complete surveys, blood draw and stool collection. Overall goals are to identify whether C. difficile is persisting in the colon mucosa after treated infection, and whether this, and other clinical and microbiome factors may be playing a role in disease recurrence.

ELIGIBILITY:
Inclusion criteria:

* Adults aged 18 and over
* Confirmed C. difficile infection based on positive C. difficile toxin PCR testing and clinical evidence of diarrhea

Exclusion criteria:

* Known pregnancy
* Prior diagnosis of C. difficile infection within 2 months of this diagnosis
* Other known active gastrointestinal infectious process
* Known diagnosis of inflammatory bowel disease, microscopic colitis, celiac disease or other inflammatory conditions
* Vulnerable adults
* Any other disease(s), condition(s) or habit(s) that would interfere with completion of study, or in the judgment of the investigator would potentially interfere with compliance to this study or would adversely affect study outcomes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients without known underlying inflammatory GI conditions with recent diagnosis and treatment of C. difficile infection, for whom the recent diagnosis was not that of recurrent disease already
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-05-05 (Actual)

PRIMARY OUTCOMES:
Mucosal presence | 1-14 days post C. Difficile treatment
  Identification of C. difficile within the colonic mucosa on stained slides from biopsy samples
Disease recurrence | 8 weeks
  Determination of recurrent C. difficile infection based on symptoms and potential clinical testing

CONTACTS AND LOCATIONS:
Overall Officials: Purna Kashyap, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials